CLINICAL TRIAL: NCT03205956
Title: Dopamine Buffering Capacity Measured by phMRI as a Novel Biomarker of Disease Progression in PD
Brief Title: Measuring Parkinson's Disease Progression
Acronym: MPDP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kevin J. Black, MD (Other)
Collaborators: The Michael J. Fox Foundation for Parkinson's Research (Unknown)
Responsible Party: Sponsor-Investigator, Kevin J. Black, MD, Professor, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 009
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; PD; levodopa
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Carbidopa

STUDY DESIGN:
Intervention Model Description: All participants receive oral carbidopa before, and i.v. levodopa during brain imaging, to measure regional cerebral blood flow responses to levodopa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PD Group (Experimental): A broad range of Parkinson's disease severity and disease duration. Some subjects will not be treated currently with levodopa, and thus likely will be early in the disease process.
  Interventions: Drug: Levodopa

INTERVENTIONS:
Drug: Levodopa — At least 1 hour after 200mg carbidopa p.o., each subject will receive an intravenous solution of levodopa in saline at a rate based on age and body mass according to the "final dose" described in Black et al 2003.The total dose for a 70-year-old, 70kg subject will be approximately 65mg.
  Subjects with untreated PD will then take 6 ± 1 weeks of clinically dosed oral carbidopa-levodopa tablets for clinical purposes and then repeat the carbidopa plus intravenous levodopa dose as above.
  Other Names: Carbidopa

SUMMARY:
The Measuring Parkinson's Disease Progression study aims to use MRI scans and a controlled dose of levodopa to find a biomarker (objective measurement) of Parkinson's disease (PD). Biomarkers would help determine the effectiveness of therapies in slowing or stopping PD progression, and accelerate the pace of research.

DETAILED DESCRIPTION:
Early in the course of Parkinson's disease, a small dose of levodopa (L-DOPA) provides benefit for many hours. The body responds as if the levodopa in the plasma filled a reservoir and then slowly leaked out to produce benefit. With disease progression, even though the same amount of levodopa circulates in the blood, the benefit wears off much faster, as if the reservoir had become leakier. This wearing off of benefit can be characterized by a single number, the effect site rate constant Ke. On average, patients with more severe disease and longer disease duration have a larger ("leakier") Ke when the response to drug is measured using clinical features like tapping speed. Unfortunately, clinical measurements are influenced by confounding factors such as patient fatigue and comfort. A direct, objective brain measure of response to levodopa may improve the reliability of this measurement. Fortunately, we can assess the effect of levodopa on the brain directly, using an MRI machine to measure blood flow in different parts of the brain. For instance, the midbrain has a robust blood flow response to a single, clinically sensible dose of levodopa. This study's goal is to validate MRI measurement of Ke in the brain as an objective, quantitative measure of disease severity in PD. We will do this by comparing MRI-based Ke values from people with PD across a wide range of disease duration and severity. In a subgroup of participants, we will do this measurement twice, once before treatment and once after 6 weeks of treatment with carbidopa-levodopa (Sinemet® and other brand names).

ELIGIBILITY:
Inclusion Criteria:

* Age 40-79 at screening
* Meet accepted diagnostic criteria for Parkinson disease

Exclusion Criteria: Key exclusion criteria:

* Deep brain stimulator (DBS)
* Pregnancy
* Patients taking a dopamine antagonist (like quetiapine) or dopamine partial agonist (like aripiprazole)
* Metal in the head or eye, or other contraindication to MRI
* Claustrophobia
* Serious neurologic disease other than PD
* Head trauma with loss of consciousness for more than 5 minutes
* Severe or unstable systemic illness
* Certain psychiatric illnesses (dementia, psychosis, current major depression)
* Current alcohol use disorder
* Subjects who feel that going without nicotine for 3-4 hours would be uncomfortable
* Currently taking an extended-release formulation of a dopamine agonist (like Mirapex ER or Requip XL)

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-19 (Actual)

PRIMARY OUTCOMES:
Ke measured by phMRI | 2 hours
  Effect site rate constant measured by serum levodopa concentrations and regional cerebral blood flow. Note, there are no outcome measures relevant to clinical care. This is not a placebo-controlled treatment study.

SECONDARY OUTCOMES:
Side effect ratings | 2 hours
  Nausea/vomiting, sleepiness, dizziness or lightheadedness, and overall feeling poorly or well, are each measured on a horizontal visual analog scale before and at the end of the i.v. levodopa infusion

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Black, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, Movement Disorders Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
We will publicly share a fully anonymized set of linked data from this study. No protected health information (PHI) will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: 36 months after completion of last participant
Access Criteria: Public
URL: https://osf.io/ezb6n/

REFERENCES:
- [Background] Black KJ, Carl JL, Hartlein JM, Warren SL, Hershey T, Perlmutter JS. Rapid intravenous loading of levodopa for human research: clinical results. J Neurosci Methods. 2003 Jul 15;127(1):19-29. doi: 10.1016/s0165-0270(03)00096-7. PMID 12865145
- [Background] Siddiqi SH, Abraham NK, Geiger CL, Karimi M, Perlmutter JS, Black KJ. The Human Experience with Intravenous Levodopa. Front Pharmacol. 2016 Jan 6;6:307. doi: 10.3389/fphar.2015.00307. eCollection 2015. PMID 26779024
- [Background] Koller JM, Vachon MJ, Bretthorst GL, Black KJ. Rapid Quantitative Pharmacodynamic Imaging with Bayesian Estimation. Front Neurosci. 2016 Apr 8;10:144. doi: 10.3389/fnins.2016.00144. eCollection 2016. PMID 27092045
- [Background] Black KJ, Acevedo HK, Koller JM. Dopamine Buffering Capacity Imaging: A Pharmacodynamic fMRI Method for Staging Parkinson Disease. Front Neurol. 2020 May 6;11:370. doi: 10.3389/fneur.2020.00370. eCollection 2020. PMID 32477245

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03205956/Prot_SAP_001.pdf